CLINICAL TRIAL: NCT01013727
Title: Functional Neuroimaging of Postural Reconstruction: Preliminary Study on a Dorsiflexion Motion of the Ankle and Comparison Between an Arm Following Postural Reconstruction Program and a Comparator Arm Following a Muscular Stretching Program
Brief Title: Functional Neuroimaging of Postural Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Basic Science
Other Study IDs: 4551
Record Dates: First submitted 2009-11-13; First posted 2009-11-16 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Healthy
Keywords: Volunteers; healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Postural Reconstruction (Experimental)
  Interventions: Radiation: SPECT : ECD-Tc99m - Neurolite, Bristol-Myers Squibb Medical Imaging
- muscular stretching (Active Comparator)
  Interventions: Radiation: SPECT : ECD-Tc99m - Neurolite, Bristol-Myers Squibb Medical Imaging

INTERVENTIONS:
Radiation: SPECT : ECD-Tc99m - Neurolite, Bristol-Myers Squibb Medical Imaging

SUMMARY:
To study in two cross-sections of healthy volunteers, with single photon emission computed tomography (SPECT), the possible changes generated in the mid-term by two rehabilitation techniques: the postural reconstruction and the muscular stretching. The changes in the cortical activation patterns will be estimated during a non-specific position of the ankle, held static.

The influence of each technique will be estimated though the evidence of a change in the functional mapping of the areas activated during the defined motor task on healthy volunteers.

DETAILED DESCRIPTION:
This is a monocentre, randomized study.

ELIGIBILITY:
Inclusion Criteria:

* male or female 18 to 35 years old

Exclusion Criteria:

* pregnant, lactating

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in the functional mapping of the areas activated during the defined motor task on healthy volunteers. | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Izzie Jacques Namer, Md, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital Strasbourg, Strasbourg, France